CLINICAL TRIAL: NCT03376113
Title: The Effect of a Brief Psychological Intervention on Reducing Self-harm Repetition: Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Academia Sinica, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201708008RINB
Record Dates: First submitted 2017-11-02; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-10

CONDITIONS: Suicide and Self-harm
Keywords: self-harm; psychological intervention
MeSH Terms: conditions — Suicide; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VHS group (Experimental): Patients will be asked to make links between critical situations and appropriate solutions in the volitional help sheet (VHS).
  Interventions: Behavioral: the volitional help sheet
- Control group (No Intervention): Patients will be asked to read the VHS. This is an active control group. That means all patients in this study will be exposed to situations and solutions in the VHS.

INTERVENTIONS:
Behavioral: the volitional help sheet — A sheet includes two columns: one shows critical situations that easily trigger self-harm; other one shows appropriate solutions for patients to prevent self-harm.
  Arms: VHS group

SUMMARY:
Recent research has focused on examining brief interventions for reducing self-harm, such as the volitional help sheet (VHS). The VHS is a theory-based psychological intervention. Two previous studies applying this tool for reducing self-harm repetition showed inconsistent results; one showed reduced subsequent self-reported suicidal ideation and behavior in patients presenting to hospital for self-harm, whilst the other showed no effect on the number of patients who re-presented to hospital with self-harm. The aim of this study is to investigate the feasibility of the VHS intervention amongst self-harm patients in Taiwan and explore its effect on self-harm repetition based on self-reported self-harm, hospital re-presentations with self-harm, and self-harm episodes from a nationwide self-harm registry. It is a two-phase study: first a qualitative study and second an exploratory randomized control trial. The first study is to interview people who self-harm about their perceptions about the VHS on the online platform, to inform the modification of VHS and the best way to intervene. The second is to examine the feasibility and effect of this intervention at the emergency department setting.

DETAILED DESCRIPTION:
Suicide is an important public health issue and leads to substantial social and economic burden. Self-harm is a significant risk factor of subsequent suicide attempt and suicide. However, previously studied interventions for reducing self-harm repetition such as long-term psychological therapies would not be feasible at acute settings such as emergency departments. It is also challenging to maintain patients who self-harm in long-term treatments. The volitional help sheet (VHS) is a brief, theory-based psychological intervention. Two recent studies applying this tool for reducing self-harm repetition showed inconsistent results; one showed reduced subsequent self-reported suicidal ideation and behavior in patients presenting to hospital for self-harm, whilst the other showed no effect on the number of patients who re-presented to hospital with self-harm. To investigate the feasibility of the VHS intervention for self-harm patients and explore its effect on self-harm repetition in Taiwan, the investigators will conduct a two-phase study: first a qualitative study and second an exploratory randomized control trial.

In phase I, the qualitative study, eight patients with recent self-harm will be recruited from the psychiatric ward and interviewed about their perceptions about the VHS and views about the best way to intervene.

In phase II, the exploratory randomized control trial, the investigators will recruit 60 patients presenting to the emergency department following an episode of self-harm. Patients will be randomly assigned (1:1) to the intervention group, which will be given the VHS intervention on an online platform, or the control group to examine the feasibility and effect of this intervention. The primary outcomes will be self-harm repetition based on: i) self-reported self-harm in a telephone based follow-up survey, ii) hospital re-presentations with self-harm based on hospital records, and iii) self-harm episodes from a nationwide self-harm registry, the National Suicide Surveillance System (NSSS). The NSSS includes a web-based reporting system and all emergency departments across the country are asked to report information about all people present to hospitals following an episode of self-harm. In addition, we will report the sub-group analyses for past self-harm hospitalisation according to the suggestion from the study testing VHS on reducing self-harm in United Kingdom.

ELIGIBILITY:
In phase I

Inclusion Criteria:

1. With self-harm experience in the past month
2. Aged 20 years or over

Exclusion Criteria:

1. With severe hallucinations or delusions or medically unfit for interview
2. Limited hands movement (e.g. seriously wounded wrists)

In phase II

Inclusion Criteria:

1. Admitted to the ER following an episode of self-harm
2. Aged 20 years or over

Exclusion Criteria:

1. With severe hallucinations or delusions or medically unfit for interview
2. Limited hands movement (e.g. seriously wounded wrists)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2017-11-03 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
The acceptability of the intervention to patients | within 6 months of study completion
  The investigators will conduct face-to-face qualitative interviews to understand the acceptability of the intervention amongst patients.
The feasibility of intervention delivery at the ER setting | within 6 months of study completion
  The investigators will conduct face-to-face qualitative interviews to understand the feasibility of intervention delivery at the ER setting.
Patient recruitment | Baseline
  Recruitment: the proportion of patients who are eligible and invited actually consent to participate.
The proportion of participating patients who can be reached by telephone contact at the 3-month follow-up. | 3 months
  The proportion of participating patients who can be reached by telephone contact at the 3-month follow-up.
The proportion of participating patients who can be reached by telephone contact at the 6-month follow-up. | 6 months
  The proportion of participating patients who can be reached by telephone contact at the 6-month follow-up.
The proportion of participating patients who can be traced from the hospital record at the 3-month. | 3 months
  The proportion of participating patients who can be traced from the hospital record at the 3-month.
The proportion of participating patients who can be traced from the hospital record at the 6-month. | 6 months
  The proportion of participating patients who can be traced from the hospital record at the 6-month.
The proportion of participating patients whose identity card number can be linked to the nationwide self-harm registry at the 6-month. | 6 months
  The proportion of participating patients whose identity card number can be linked to the nationwide self-harm registry at the 6-month.
The proportion of participating patients whose identity card number can be linked to the nationwide self-harm registry at the 3-month. | 3 months
  The proportion of participating patients whose identity card number can be linked to the nationwide self-harm registry at the 3-month.
Change in scores on a self-report suicidal behaviors assessment from baseline to 3 months | Baseline, 3 months
  As measured by the total score of the Suicidal Behaviors Questionnaire-Revised (SBQ-R), a 4-item scale for assessing suicidal behavior and ideation. The total score ranges from 3 to 18.
Change in scores on a self-report suicidal behaviors assessment from baseline to 6 months | Baseline, 6 months
  As measured by the total score of the Suicidal Behaviors Questionnaire-Revised (SBQ-R), a 4-item scale for assessing suicidal behavior and ideation. The total score ranges from 3 to 18.
Number of repeat self-harm episodes per person in 3 months after intervention based on hospital records | 3 months
  Number of repeat self-harm episodes per person in 3 months after intervention based on hospital records
Number of repeat self-harm episodes per person in 3 months after intervention recorded in the nationwide self-harm registry | 3 months
  Number of repeat self-harm episodes per person in 3 months after intervention recorded in the nationwide self-harm registry
Number of repeat self-harm episodes per person in 6 months after intervention based on hospital records | 6 months
  Number of repeat self-harm episodes per person in 6 months after intervention based on hospital records
Number of repeat self-harm episodes per person in 6 months after intervention recorded in the nationwide self-harm registry | 6 months
  Number of repeat self-harm episodes per person in 6 months after intervention recorded in the nationwide self-harm registry
Time to next self-harm repetition (in days) following randomization | 6 months
  Time to next self-harm repetition (in days) following randomization according to hospital records and a nationwide self-harm registry.

SECONDARY OUTCOMES:
Times of use of the volitional help sheet | 6 months
  Times of use of the volitional help sheet based on the number of visits to the individualized website of the volitional help sheet.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Sen Chang, MD, MSc, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793